CLINICAL TRIAL: NCT05274997
Title: A Single-arm, Phase II Study to Evaluate the Efficacy and Safety of Linperlisib (YY-20394) Monotherapy in Patients With Relapsed or Refractory Peripheral T/NK Cell Lymphoma
Brief Title: A Phase II Study of Linperlisib (YY-20394) in Patients With Relapsed or Refractory Peripheral T/NK Cell Lymphoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shanghai YingLi Pharmaceutical Co. Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: YY-20394-012
Record Dates: First submitted 2022-02-23; First posted 2022-03-11 (Actual); Last update posted 2022-10-21 (Actual); Status verified 2022-02

CONDITIONS: Peripheral T/NK Cell Lymphoma (R/R PTCL)

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- YY-20394 (Experimental): Administer linperlisib (YY-20394) 80 mg (4 tablets) orally with water, once daily, in a 28-day cycle.
  Interventions: Drug: YY-20394

INTERVENTIONS:
Drug: YY-20394 — Linperlisib is a strong and selective small-molecule PI3K-δ (a protein involves in the survival of cells) inhibitor, which is able to interfere with the growth, migration and survival of T/NK lymphoma cells.
  Other Names: Linperlisib

SUMMARY:
This is a Phase II, single-arm study to evaluate the efficacy, safety, and PK of oral linperlisib (YY-20394) monotherapy in adult patients with R/R Peripheral T/NK Cell Lymphoma. The study will be conducted at approximately 15 sites in United States.

ELIGIBILITY:
Inclusion Criteria:

1. Adult patient ≥18 years of age at the time of signing the informed consent.
2. Diagnosis of one of the following histologic subtypes of PTCL, pathologically confirmed, as defined by the WHO 2017 classification system:

   1. Peripheral T-cell lymphoma-not otherwise specified (PTCL-NOS)
   2. Angioimmunoblastic T-cell lymphomas (AITL)
   3. Anaplastic large cell lymphoma (ALCL). ALK positive or ALK negative
   4. Natural-killer/T-cell lymphoma (NKTCL)
   5. Monomorphic epitheliotropic intestinal T-cell lymphoma (MEITL).
3. Has received and failed at least one line of systemic therapy.
4. Not a candidate for autologous or allogeneic transplantation.
5. For patients with CD30+ PTCL, progressed on or are ineligible or intolerant to brentuximab vedotin.
6. Agree to provide archived tumor tissue samples or undergo pretreatment fresh tissue biopsy.
7. Has radiographically measurable disease as per Lugano Criteria with at least one measurable disease lesion > 1.5 cm in at least one dimension (which has not been previous radiated) by 18FDG-PET-CT, MRI, or diagnostic CT within 28 days prior to start of study treatment.
8. Has an Eastern Cooperative Oncology Group (ECOG) performance status of 0 to 1.
9. Has adequate organ function as defined below:

   System Laboratory Value Haematological Absolute neutrophil count
   * 1.0×109/L Note: No growth factor supports within 14 days of first dose Platelet count
   * 75×109/L Note: ≥50 × 109/L for patients with bone marrow infiltration No blood product transfusion is allowed within 14 days of first dose. Haemoglobin
   * 8.0 g/L Note: criteria must be met without erythropoietin dependency and no blood product transfusion is allowed within 14 days of first dose Hepatic Total bilirubin

     * 1.5×ULN Note: Patients with Gilbert's Syndrome or other benign congenital hyperbilirubinemia may be eligible at the Investigator's discretion in consultation with the Medical Monitor, if ≤ 3 × ULN Alanine aminotransferase
     * 2.5×ULN Note: ≤ 5 × ULN if there is liver involvement by lymphoma Aspartate aminotransferase
     * 2.5×ULN Note: ≤ 5 × ULN if there is liver involvement by lymphoma Renal CrCl calculated by Cockcroft-Gault formula CrCl ≥50 mL/min Coagulation INR < 1.5 without anti-coagulation therapy Activated partial thromboplastin time aPTT ≤1.5 ULN Cardiac Left ventricular ejection fraction LVEF ≥ 50% by an echocardiogram (ECHO) or multigated acquisition scan (MUGA). QTcF <470 ms Abbreviations: CrCl=creatinine clearance; RBC=red blood cell; QTcF=QT interval corrected using Fridericia's formula; ULN=upper limit of normal.
10. Male patients are eligible to participate if they agree to use a highly effective contraception as detailed in Appendix 4 of this protocol during the treatment period and for at least 3 months after the last dose of study treatment and refrain from donating sperm during this period. 11. Female patients are eligible to participate if they are not pregnant (see Appendix 4), not breastfeeding, and at least one of the following conditions applies:

    * Not a woman of childbearing potential (WOCBP) as defined in Appendix 4. OR
    * A WOCBP who agrees to use a contraceptive method that is highly effective (with a failure rate of <1% per year), or be abstinent from heterosexual intercourse as their preferred method and usual lifestyle as described in Appendix 4, beginning the time of informed consent, during the treatment period and for at least 3 months after the last dose of study treatment.

A WOCBP must have a negative serum pregnancy within 72 hours of the first dose of study treatment.

12. Patient is capable of giving signed informed consent. 13. Must be willing and able to adhere to the study and lifestyle restrictions as judged by the investigator.

Exclusion Criteria:

* 1. Patients with peripheral T-cell lymphoma having known central nervous system (CNS) invasion (either CNS lymphoma or leptomeningeal lymphoma).

  2. Has clinically significant (i.e., active) cardiovascular disease: cerebral vascular accident/stroke (<6 months prior to enrollment), myocardial infarction (<6 months prior to enrollment), unstable angina, congestive heart failure (New York Heart Association Classification Class ≥II), or serious cardiac arrhythmia requiring medication, any other cardiac disorder not suitable for participation in this study based on the judgment of the investigator. Note: During the treatment period, patients should not take medication that may prolong the QT (such as antiarrhythmic drugs).

  3. Presence of multiple factors affecting drug administration and absorption such as inability to swallow, diarrhea of CTCAE Grade >1, and ileus.

  4. Has a history of or concurrent interstitial lung disease of any severity and/or severely impaired lung function.

  5. Prior history of drug-induced colitis or drug-induced pneumonitis. 6. Has active viral, bacterial, fungal infection or other serious infection requiring systemic treatment within 14 days before the first dose of study treatment. Routine antimicrobial prophylaxis is permitted.

  7. Medical history of active bleeding within 2 months prior to study entry, or susceptible to bleeding by the judgement of investigator.

  8. Use of therapeutic doses of warfarin sodium (Coumadin), or any other coumarin-derivative anticoagulants. The administration of low-molecular weight heparin is allowed.

  9. Unresolved toxicities from prior anti-tumor therapy, defined as not having resolved to CTCAE version 5.0 grade 0 or 1 with the exception of alopecia and peripheral neuropathy.

  10. Medical history of other primary malignant tumors in the past 5 years, or any evidence of residual disease from a previously diagnosed malignancy. Note: Exceptions are patients with basal cell carcinoma of the skin, squamous cell carcinoma of the skin or carcinoma in situ (e.g., breast, cervical cancer in situ, superficial bladder tumors [Ta and Tis; carcinoma in situ]) who have undergone curative therapy with no evidence of recurrence, localized prostate cancer previously fully resected undergoing surveillance or other adequately treated Stage 1 cancer currently in complete remission.

  11. Has received prior treatment with linperlisib (YY-20394), or other PIK3-δ inhibitors. Patients who have received prior treatment with other PIK3-δ inhibitors, but were intolerant to them, maybe included.

  12. Has received prior treatment with rituximab or other unconjugated antibody treatment within 28 days (21 days if clear evidence of progressive disease or immediate treatment is mandated) prior to the first dose of study treatment.

  13. Has received radioimmunoconjugates or toxin conjugates within 12 weeks before the first dose of study treatment.

  14. Has had received prior systemic anticancer therapy, or definitive radiotherapy ≤28 days (14 days for palliative radiation) prior to the first dose of study treatment.

  15. Has received prior targeted small molecule therapy ≤14 days or 5 half-lives whichever is longer.

  16. Has undergone major surgery (excluding lymph node biopsy) or significant trauma ≤4 weeks before the first dose of study treatment. Note: patients must have recovered adequately from surgery prior to starting study treatment.

  17. Use of medications or foods that are strong cytochrome CYP3A inhibitors, strong CYP3A inducers within 14 days prior to first dose of study treatment or 5 half-lives of the given drug, whichever is longer.

  18. Use of any drug that may result in QT prolongation (e.g., antiarrhythmic agents) cannot be interrupted during the study.

  19. Has a history of immunodeficiency or autoimmune disease has received systemic steroids (in dosing exceeding 10 mg daily of prednisolone equivalent) or any other form of immunosuppressive therapy within 7 days of the first dose of study treatment. The use of physiological doses of corticosteroids may be approved after consultation with the Medical Monitor.

  20. Has received a live vaccination within 30 days before the first dose of study treatment or is scheduled to be administered during the study period. Examples of live vaccines include but are not limited to the following: measles, mumps, rubella, varicella/zoster, yellow fever, Bacille Calmette-Guérin (BCG) and typhoid vaccine. Seasonal influenza vaccines for injection are generally killed virus vaccines and are allowed; however, intranasal influenza vaccines (e.g., FluMist®) are live attenuated vaccines and are not allowed.

  21. Human immunodeficiency virus (HIV) infection with a current or a known history of acquired immunodeficiency syndrome (AIDS)-defining illness or HIV infection with a CD4+ T cell count <350 cells/μL and an HIV viral load more than 400 copies/μL.

  22. Patients with active viral (any etiology) hepatitis are excluded. Patients with a history of hepatitis C virus (HCV) infection who have completed curative antiviral treatment and have a viral load below the limit of quantification may be eligible and should be discussed with the Medical Monitor.

  23. Patients who have a positive PCR test for CMV at screening will not be enrolled in the study.

  24. Has a history or current evidence of any condition, laboratory abnormality or other circumstances that might confound the results of the study or interfere with participation for the full duration of the study, such that it is not in the best interests of the patient to take part in the study.

  25. Patient is pregnant or breastfeeding or expecting to conceive of father children for the duration of the study.

  26. Has a history of hypersensitivity to linperlisib (YY-20394) and/or any excipients.

  27. Has a known psychiatric disorder that would interfere with compliance with the requirements of the study.

  28. Is a regular user of illicit or recreational drugs or has a recent history (within the last year) of drug or alcohol abuse or dependence.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 97 (Estimated)
Dates: Start 2022-05-01 (Actual); Primary Completion 2023-01-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
overall response rate (ORR) | Throughout the study for approximately 2 years
  Overall response rate (ORR = CR + PR), from start of treatment to first documented response, measured by Lugano 2014 Response Criteria for NHL (Cheson 2014)

SECONDARY OUTCOMES:
duration of response (DOR) | Throughout the study for approximately 2 years
  DOR, defined as time from first documentation of a response (PR or CR) to the first documented disease progression or death due to any cause, whichever occurs first, for those patients with a PR or CR.
progression-free survival (PFS), | Throughout the study for approximately 2 years
  PFS, defined as the time from start of treatment to first documented disease progression or death due to any cause, whichever occurs first.
Overall survival (OS) | Throughout the study for approximately 2 years
Time to response (TTR) | Throughout the study for approximately 2 years
AE | Throughout the study for approximately 2 years
  Incidence of Adverse events (AEs) using the National Cancer Institute Common Terminology Criteria for Adverse Events (NCI-CTCAE) Version 5.0
AUClast | Throughout the study for approximately 2 years
  PK parameters
AUCinf | Throughout the study for approximately 2 years
  PK parameters
Cmin | Throughout the study for approximately 2 years
  PK parameters
Cmax | Throughout the study for approximately 2 years
  PK parameters
T1/2 | Throughout the study for approximately 2 years
  PK parameters
Tmax | Throughout the study for approximately 2 years
  PK parameters

CONTACTS AND LOCATIONS:
Overall Officials: Ranjit Nair, MD., Principal Investigator — MD Anderson, Houston TX 77030 Study Chair: Swaminathan P Iyer MD
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

IPD SHARING:
Plan to Share IPD: No